CLINICAL TRIAL: NCT04935645
Title: The Effect of Progressive Muscle Relaxation on Abdominal Pain and Distension in Colonoscopy Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mardin Artuklu University (Other)
Responsible Party: Principal Investigator, Seher Tanrıverdi, Research asistant, Mardin Artuklu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Mardin Artuklu University
Record Dates: First submitted 2021-05-25; First posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Abdominal Pain
Keywords: Colonoscopy; Abdominal Pain; Nursing; relaxation; exercise
MeSH Terms: conditions — Abdominal Pain; Motor Activity | interventions — Autogenic Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The experimental group was informed about progressive muscle relaxation (PMR) before colonoscopy. PMR audio recordings were given to the patients. Abdominal pain and distention scores were determined after colonoscopy. PMR was applied to the patients for 30 minutes. These scores were determined again after exercise and at the 2nd, 4th, 8th, 12th, 16th, and 24th hours.
  Interventions: Behavioral: Progressive Muscle Relaxation
- Control Group (No Intervention): VAS pain and VAS distension scores of the control group were determined after colonoscopy and 30 minutes later. VAS form was given to all patients to determine VAS abdominal pain and VAS distension scores at the 2nd, 4th, 8th, 12th, 16th and 24th hours after the procedure. The day after the colonoscopy, post test data were collected.

INTERVENTIONS:
Behavioral: Progressive Muscle Relaxation — PMR is a technique that provides relaxation in the whole body by voluntary and regular relaxation of large muscle groups in the human body, which is included in mind-body applications.
  Arms: Experimental Group

SUMMARY:
Patients undergoing colonoscopy were divided into progressive relaxation exercises and control groups. Pretest and posttest abdominal pain and distention scores of the patients were determined after colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing colonoscopy
* Those who do not have communication problems,
* After the colonoscopy procedure, the abdominal pain score is evaluated by VAS and is 4 or higher,
* Evaluation of the distension score of 4 and above with VAS after the colonoscopy procedure,
* Be 18 years old or older.

Exclusion Criteria:

* Being a hospitalized patient undergoing colonoscopy,
* Be younger than 18 years old
* To have used complementary and alternative methods during the research,
* Any physical problem that may prevent you from doing the exercises,
* Having a cognitive illness
* Refusing to participate in the research,
* Failing to complete surveys.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Individual Introductory Information Form | 15 minutes
  This form, which was created by the researcher with the support of the relevant literature, consists of 11 questions questioning the patients' education level, age,gender, employment status, marital status,income level, the coping methods they use when there is distension in their daily lives, the coping methods they use when there is pain in their daily lives, the status of having a colonoscopy before, the history of abdominal pain and distension of those who have a colonoscopy experience.

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) | 10 minutes
  The patient was asked to make a mark on a 10 cm horizontal line on the Visual analog scale showing his current state. In this study, for pain and distension; Markings were made on a 10 cm horizontal line, one end of which indicates that the patient's pain is very good (0 = no pain) and the other end is that the patient's pain is very bad (10 = most severe). The distance from the point where there was no pain and distension (0) to the point marked by the patient was measured. The value found shows the severity of pain and distention of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Seher Tanrıverdi, Principal Investigator — Mardin Artuklu University
Locations (1):
- Mardin State Hospital, Mardin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
can be reviewed by other researchers after the study has been published.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: data will be shared as long as they are published
Access Criteria: publication page

REFERENCES:
- [Background] Levy I, Gralnek IM. Complications of diagnostic colonoscopy, upper endoscopy, and enteroscopy. Best Pract Res Clin Gastroenterol. 2016 Oct;30(5):705-718. doi: 10.1016/j.bpg.2016.09.005. Epub 2016 Sep 14. PMID 27931631
- [Background] Pan CX, Morrison RS, Ness J, Fugh-Berman A, Leipzig RM. Complementary and alternative medicine in the management of pain, dyspnea, and nausea and vomiting near the end of life. A systematic review. J Pain Symptom Manage. 2000 Nov;20(5):374-87. doi: 10.1016/s0885-3924(00)00190-1. PMID 11068159
- [Background] Park DI, Kim HJ, Park JH, Cho YK, Sohn CI, Jeon WK, Kim BI, Ryu SH, Sung IK. Factors affecting abdominal pain during colonoscopy. Eur J Gastroenterol Hepatol. 2007 Aug;19(8):695-9. doi: 10.1097/01.meg.0000219097.32811.24. PMID 17625440
- [Background] Steffenssen MW, Al-Najami I, Baatrup G. Patient-reported minor adverse events after colonoscopy: a systematic review. Acta Oncol. 2019;58(sup1):S22-S28. doi: 10.1080/0284186X.2019.1574979. Epub 2019 Feb 20. PMID 30784355
- [Result] Lahmann C, Rohricht F, Sauer N, Noll-Hussong M, Ronel J, Henrich G, von Arnim A, Loew T. Functional relaxation as complementary therapy in irritable bowel syndrome: a randomized, controlled clinical trial. J Altern Complement Med. 2010 Jan;16(1):47-52. doi: 10.1089/acm.2009.0084. PMID 20064018